CLINICAL TRIAL: NCT04100928
Title: Evaluating the Well-being Among Dental Students With Warwick-Edinburg Mental Well-Being Scale and the Relationship Between Mental Well-being and Socio-demographic Findings
Brief Title: Evaluating the Well-being Among Dental Students With Warwick-Edinburg Mental Well-Being Scale
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, asistant professor, Baskent University
Other Study IDs: BaskentU6
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Well Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dental students — WEMWBS and a questionnaire included demographic details and social background, lifestyle behaviors was applied to the participants.
  Other Names: no intervention was made

SUMMARY:
The present study was conducted to measure the mental well-being amongst dental students by using Warwick-Edinburg Mental Well-being Scale (WEMWBS) and investigate factors affecting well-being among dental students.

DETAILED DESCRIPTION:
The survey schedule was planned to be independent of the students' assessment period and the questionnaire was administered to the students when they were attending a lecture together. After the lecture, a researcher explained to the students the purpose of this survey and assured them of confidentiality. Participation in this study was also voluntary, and all participants remained anonymous. The questionnaire was given to all participants after explaining the purpose of the study. The questionnaire included demographic details (age, gender, year of study), social background (parents' education levels, family income, first choice for admission, living accommodation) and lifestyle behaviors (smoking status, presence of regular sport activity and hobby). In addition, Warwick-Edinburg Mental Well-Being Scale was applied to the participants of this study.

ELIGIBILITY:
Inclusion Criteria:

to be officially registered in the faculty of dentistry, Baskent University

Exclusion Criteria:

unwilling to participate

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All students in the faculty of dentistry, Baskent University
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburg Mental Well-being Scale | day 1
  Individuals completing the scale are required to tick the box that best describes their experience of each statement over the past two weeks using a 5-point Likert scale (none of the time, rarely, some of the time, often, all of the time). The Likert scale represents a score for each item from 1 to 5 respectively, giving a minimum score of 14 and maximum score of 70.

CONTACTS AND LOCATIONS:
Overall Officials: yasemin sezgin, Study Director — Dr.
Locations (1):
- Yasemin Sezgin, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided